CLINICAL TRIAL: NCT07242456
Title: Head-to-head Comparison of Tegoprazan 50 mg BID Plus Amoxicillin 1 g TID Versus Vonoprazan 20 mg BID Plus Amoxicillin 1 g TID for Helicobacter Pylori Eradication: A Randomized, Open-label, Parallel-group Study
Brief Title: Head-to-head Study of Tegoprazan 50 mg BID Plus Amoxicillin 1 g TID vs. Vonoprazan 20 mg BID Plus Amoxicillin 1 g TID for H. Pylori Eradication
Acronym: TV-HP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, shenhongzhang, Associate Chief Physician, Department of Gastroenterology, Hangzhou First People's Hospital, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV-HP-2024-01; BCF-LX-XH-20221014-26 (Other Grant/Funding Number: Bethune Charitable Foundation)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-01

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan; Amoxicillin; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two treatment arms and will receive the assigned regimen for 14 days. Both groups will be followed in parallel, with no crossover or sequence changes. Outcomes will be assessed at predefined follow-up visits.
Masking Description: Not applicable. This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan + Amoxicillin (14-day dual therapy) (Experimental): Participants in this arm will receive tegoprazan 50 mg taken orally twice daily and amoxicillin 1 g taken orally three times daily for 14 consecutive days. All medications are administered with water after meals. Participants will be followed for assessment of H. pylori eradication 4 to 8 weeks after completing treatment.
  Interventions: Drug: Tegoprazan; Drug: Amoxicillin
- Vonoprazan + Amoxicillin (14-day dual therapy) (Experimental): Participants in this arm will receive vonoprazan 20 mg taken orally twice daily and amoxicillin 1 g taken orally three times daily for 14 consecutive days. All medications are administered with water after meals. Participants will be followed for assessment of H. pylori eradication 4 to 8 weeks after completing treatment.
  Interventions: Drug: Amoxicillin; Drug: Vonoprazan

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg orally twice daily for 14 days.
  Arms: Tegoprazan + Amoxicillin (14-day dual therapy)
Drug: Amoxicillin — Amoxicillin 1 g orally three times daily for 14 days.
Drug: Vonoprazan — Vonoprazan 20 mg orally twice daily for 14 days.
  Arms: Vonoprazan + Amoxicillin (14-day dual therapy)

SUMMARY:
This study is a randomized, open-label, parallel-group clinical trial designed to compare two 14-day dual therapies for the eradication of Helicobacter pylori (H. pylori) infection. Participants will be randomly assigned to receive either tegoprazan 50 mg twice daily plus amoxicillin 1 g three times daily, or vonoprazan 20 mg twice daily plus amoxicillin 1 g three times daily.

The primary purpose of this study is to evaluate whether the tegoprazan-based regimen is non-inferior to the vonoprazan-based regimen in terms of H. pylori eradication rates. Eradication will be assessed 4 to 8 weeks after completing therapy using a ^13C-urea breath test. Secondary objectives include assessing treatment-related adverse events, tolerability, and medication adherence.

This study involves adult participants with confirmed H. pylori infection. All study medications are orally administered, and both regimens use drugs with well-established safety profiles. The study is investigator-initiated and conducted at Hangzhou First People's Hospital.

DETAILED DESCRIPTION:
This investigator-initiated, randomized, open-label, parallel-group study is designed to compare two potassium-competitive acid blocker (P-CAB)-based dual therapies for the eradication of Helicobacter pylori (H. pylori) infection. The study evaluates a 14-day regimen of tegoprazan 50 mg twice daily combined with amoxicillin 1 g three times daily versus a 14-day regimen of vonoprazan 20 mg twice daily combined with amoxicillin 1 g three times daily.

H. pylori infection is a major cause of chronic gastritis, peptic ulcer disease, and gastric cancer. Rising antimicrobial resistance and variable acid suppression with conventional proton pump inhibitors (PPIs) have highlighted the need for alternative treatment strategies. P-CABs, including tegoprazan and vonoprazan, provide rapid, potent, and sustained acid suppression and may enhance the efficacy of high-dose amoxicillin dual therapy. Despite their increasing clinical use, head-to-head comparative evidence between different P-CAB-based dual therapies is limited.

The primary objective of this study is to determine whether the tegoprazan-based dual regimen is non-inferior to the vonoprazan-based dual regimen in terms of H. pylori eradication rate, assessed by a ^13C-urea breath test performed 4 to 8 weeks after treatment completion. Secondary assessments include treatment-emergent adverse events, serious adverse events, gastrointestinal symptom changes, and medication adherence.

Eligible participants are adults with confirmed H. pylori infection who have not received recent eradication therapy or antibiotics with anti-H. pylori activity. The study drugs have established safety profiles and are administered orally. Participants will be randomized in a 1:1 ratio and followed until completion of eradication testing and safety assessments. Data will be analyzed using both intention-to-treat and per-protocol populations.

This study is conducted at Hangzhou First People's Hospital and is intended to provide direct comparative data to guide the selection of P-CAB-based dual therapy regimens in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 18 to 70 years. 2. Confirmed Helicobacter pylori infection based on at least one positive test (13C-urea breath test, rapid urease test, histology, or stool antigen test). 3. Able and willing to provide written informed consent. 4. Able to comply with study procedures and visits. 5. For females of childbearing potential: agreement to use effective contraception during the study period.

Exclusion Criteria:

* 1. Previous Helicobacter pylori eradication therapy within the past 12 months. 2. Use of antibiotics, bismuth compounds, or other medications with anti-H. pylori activity within 4 weeks before baseline testing. 3. Use of proton pump inhibitors, P-CABs, or H2-receptor antagonists within 2 weeks before baseline testing. 4. Known allergy or intolerance to tegoprazan, vonoprazan, amoxicillin, or any beta-lactam antibiotic. 5. Known severe hepatic impairment (e.g., Child-Pugh C) or severe renal impairment (e.g., eGFR < 30 mL/min/1.73 m²). 6. History of gastric surgery (except minor endoscopic procedures that do not affect gastric anatomy).

  7. Active gastrointestinal bleeding or suspected gastric malignancy. 8. Pregnant or breastfeeding women. 9. Participation in another interventional clinical trial within the past 30 days.

  10. Any medical or psychiatric condition that, in the investigator's judgment, could interfere with study participation or pose unacceptable risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori Eradication Rate (ITT and PP) | 4 to 8 weeks after completion of the 14-day treatment regimen
  H. pylori eradication will be defined as a negative ^13C-urea breath test performed at the follow-up visit. Eradication rates will be assessed in both the intention-to-treat (ITT) and per-protocol (PP) populations. A participant will be considered eradicated only if the test result is negative without the use of prohibited medications.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose to 2 weeks after completion of treatment (approximately 4 weeks total)
  Number and proportion of participants experiencing at least one treatment-emergent adverse event, classified by severity and relationship to study medication.
Incidence of Serious Adverse Events (SAEs) | From first dose to end of study follow-up (up to 10 weeks)
  Number and proportion of participants experiencing at least one serious adverse event, as defined by international regulatory criteria.
Rate of Treatment Discontinuation Due to Adverse Events | During the 14-day treatment period
  Proportion of participants who permanently discontinue the study medication because of adverse events.
Change in Gastrointestinal Symptom Scores | Baseline to end of 14-day treatment
  Change from baseline in gastrointestinal symptom scores (e.g., nausea, bloating, abdominal pain), measured using a standardized symptom questionnaire.
Medication Adherence Rate | During the 14-day treatment period
  Percentage of prescribed doses taken by participants, assessed using pill counts and/or patient diaries.

OTHER OUTCOMES:
Subgroup Analysis by CYP2C19 Metabolizer Status | At the time of primary eradication assessment (4 to 8 weeks after completion of the 14-day treatment regimen)
  If genotyping is performed, participants will be categorized into metabolizer groups (e.g., poor, intermediate, extensive, rapid metabolizers). H. pylori eradication rates will be compared across CYP2C19 phenotypes to explore potential differences in treatment response to P-CAB-based dual therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Department of Gastroenterology (Helicobacter pylori Standardized Diagnosis and Treatment Clinic, National Demonstration Center), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This study is a single-center, investigator-initiated clinical trial, and there is no plan to make de-identified IPD available to external researchers. Summary results will be published in peer-reviewed journals.